CLINICAL TRIAL: NCT02045524
Title: A Pilot Single Dose Crossover Pharmacokinetics Study Of JDP-205 Injection, 10 mg, In Healthy Male And Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: JDP Therapeutics, Inc. (Industry)
Collaborators: Algorithme Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ETTAU-01P (CTN-P1-571)
Record Dates: First submitted 2014-01-22; First posted 2014-01-27 (Estimated); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Acute Urticaria

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Injection location1 (Experimental): Single dose IM injection
  Interventions: Other: Deep muscle injection
- Injection location 2 (Experimental): Single dose IM Injection
  Interventions: Other: Sub-Q Injection

INTERVENTIONS:
Other: Deep muscle injection
  Arms: Injection location1
Other: Sub-Q Injection
  Arms: Injection location 2

SUMMARY:
The objective of this study was to investigate the pharmacokinetics (PK) of JDP-205 injection at 10 mg dose administered by intramuscular injection using various injection techniques in healthy male and female volunteers after a single dose administration.

ELIGIBILITY:
Inclusion Criteria:

Volunteers meeting all of the following criteria were considered for enrollment in the study:

1. Male or female volunteer
2. Volunteer aged of at least 18 years
3. Volunteer with a body mass index (BMI) greater than or equal to 18.50 and below 30.00 kg/m2
4. Non- or ex-smokers; an ex-smoker being defined as someone who completely stopped smoking for at least 12 months before day 1 of this study.
5. Availability for the entire study period
6. Motivated volunteer and absence of intellectual problems likely to limit the validity of consent to participate in the study or the compliance with protocol requirements; ability to cooperate adequately; ability to understand and observe the instructions of the physician or designee
7. Clinical laboratory values within the laboratory's stated normal range; if not within this range, they must be without any clinical significance
8. Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings on physical examination (including the examination of the anterolateral thigh muscles) and/or clinical laboratory evaluations (hematology, biochemistry, ECG and urinalysis)
9. Willingness to adhere to the protocol requirements as evidenced by the informed consent form (ICF) duly read, signed and dated by the volunteer

Exclusion Criteria:

Volunteers presenting any of the following were not included in the study:

1. Females who are pregnant or are lactating
2. Females of childbearing potential who refuse to use an acceptable contraceptive regimen throughout the entire duration of the study (from the screening visit until study completion)
3. History of significant hypersensitivity to cetirizine or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs
4. Presence of significant gastrointestinal, liver or kidney disease, or any other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs or known to potentiate or predispose to undesired effects
5. History of significant gastrointestinal, liver or kidney disease that may affect drug bioavailability
6. Presence of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic or dermatologic disease
7. Suicidal tendency, history of or disposition to seizures, state of confusion, clinically relevant psychiatric diseases
8. Presence of out-of-range cardiac interval (PR < 110 msec, PR > 200 msec, QRS < 60 msec, QRS >110 msec and QTc > 440 msec) on the screening ECG or other clinically significant ECG abnormalities
9. Known presence of rare hereditary problems of galactose and /or lactose intolerance
10. Maintenance therapy with any drug, or significant history of drug dependency or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
11. Any clinically significant illness in the previous 28 days before day 1 of this study
12. Use of any enzyme-modifying drugs, including strong inhibitors of cytochrome P450 (CYP) enzymes (such as cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem and HIV antivirals) and strong inducers of CYP enzymes (such as barbiturates, carbamazepine, glucocorticoids, phenytoin, rifampin and St John's Wort), in the previous 28 days before day 1 of this study
13. Use of antihistaminic medication in the previous 7 days before day 1 of this study
14. Any history of tuberculosis and/or prophylaxis for tuberculosis
15. Positive urine screening of ethanol and/or drugs of abuse
16. Positive results to HIV, HBsAg or anti-HCV tests
17. Females who are pregnant according to a positive serum pregnancy test
18. Volunteers who took an Investigational Product (in another clinical trial) or donated 50 mL or more of blood in the previous 28 days before day 1 of this study
19. Donation of 500 mL or more of blood (Canadian Blood Services, Hema-Quebec, clinical studies, etc.) in the previous 56 days before day 1 of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Difference in pharmacokinetics: Difference in AUC | 8 hours post dose
Differences in pharmacokinetics: difference in Cmax | 8 hours post dose

CONTACTS AND LOCATIONS:
Locations (1):
- Algorithme Pharma, Montreal, Quebec, Canada